CLINICAL TRIAL: NCT04654884
Title: Auricular Acupuncture as an add-on Treatment for Symptoms of Anxiety Within Affective Out-patient Care
Brief Title: Auricular Acupuncture as an add-on Treatment for Symptoms of Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-06078 B
Record Dates: First submitted 2020-11-03; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Anxiety Disorders; Post Traumatic Stress Syndrome
MeSH Terms: conditions — Anxiety Disorders; Combat Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: Randomisation into two groups. Group 1 will receive AA as an adjunctive therapy to TaU (i.e. individual counseling therapy, psycho therapy, pharmacological therapy)Group 2, the control group, will receive TaU.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): The participants in group 1 will receive AA as an adjunctive therapy to TaU (i.e. individual counseling therapy, psycho therapy, pharmacological therapy) during 8 weeks.
  Interventions: Other: Auricular acupuncture (AA)
- Group 2 (No Intervention): Group 2, the control group, will receive TaU and will, just like goup 1, have a follow-up after 8 weeks.

INTERVENTIONS:
Other: Auricular acupuncture (AA) — The add-on treatment will be administered at the treatment sessions with their caregiver (i.e. registered nurse, psychologist, curator), and at each session the participants receive 5 sterile stainless needles in each outer ear. The needling is standardised according to the NADA-protocol. The needles will remain in the outer ears for approximately 45 minutes, and will be removed by the care giver.
  Arms: Group 1

SUMMARY:
Mental illness is very common in todays' society, and it is the most common cause for sick leave in Sweden. Affective diseases, such as different states of anxiety and depression, are the two most common conditions of mental illness that has been reported by different workplaces in Sweden. Pharmacological treatment of anxiety using benzodiazepines, tends to be long, and it may lead to substance dependence, as well as severe side effects such as increased anxiety levels, cognitive impact and psychomotor effects. The Swedish Council on Health Technology Assessment (SBU) have identified that there are scientific knowledge gaps that needs to be filled regarding the mental illness care, such as anxiety. There is a need for evaluations of non-pharmacological, complementary treatments as well as research with a high methodological quality.

Acupuncture is a nonpharmacological treatment method based on complementary medicine, for which interest has increased over the last years. It has, to some extent, been introduced in the ordinary health care system. Auricular acupuncture (AA) is a branch of acupuncture where needles are inserted in different areas in the outer ears AA has been used to treat anxiety as well as vid depression and post-traumatic stress syndrome (PTSD) among veterans. A standardised insertion pattern, defined as the National Acupuncture Detoxification Association (NADA) protocol, is normally practised, and it has also been used to treat insomnia. Evaluations has shown that AA according to the NADA-protocol has a calming effect and seem to alleviate symptoms of anxiety, depression and to some extent, also sleeping difficulties. The aim of this study is to study and evaluate effects of AA as an add-on treatment to treatment as usual (TaU) within affective outpatient care for patients suffering from symptoms of anxiety and depression.

A prospective, non-inferiority randomised controlled study (RCT) with a number of (N=72) participants will be conducted to answer the study aims. A qualitative interview study will also be conducted to find out how the patients experience AA as an adjunctive therapy.

DETAILED DESCRIPTION:
Mental illness is very common in todays' society, and it is the most common cause for sick leave in Sweden. Affective diseases, such as different states of anxiety and depression, are the two most common conditions of mental illness that has been reported by different workplaces in Sweden. Pharmacological treatment of anxiety using benzodiazepines, tends to be long, and it may lead to substance dependence, as well as severe side effects such as increased anxiety levels, cognitive impact and psychomotor effects. The Swedish Council on Health Technology Assessment (SBU) have identified that there are scientific knowledge gaps that needs to be filled regarding the mental illness care, such as anxiety. There is a need for evaluations of non-pharmacological, complementary treatments as well as research with a high methodological quality.

Acupuncture is a nonpharmacological treatment method based on complementary medicine, for which interest has increased over the last years. It has, to some extent, been introduced in the ordinary health care system. Auricular acupuncture (AA) is a branch of acupuncture where needles are inserted in different areas in the outer ears AA has been used to treat anxiety as well as vid depression and post-traumatic stress syndrome (PTSD) among veterans. A standardised insertion pattern, defined as the National Acupuncture Detoxification Association (NADA) protocol, is normally practised, and it has also been used to treat insomnia.

Evaluations has shown that AA according to the NADA-protocol has a calming effect and seem to alleviate symptoms of anxiety, depression and to some extent, also sleeping difficulties.

The aim of this study is to study and evaluate effects of AA as an add-on treatment to treatment as usual (TaU) within affective outpatient care.

regarding:

* Anxiety/depression: is the treatment symptom relieving?
* Does it change the participants' intake addictive drugs (i.e. benzodiazepines)?
* Sleep: Is there some improvement in any sleep disorders that are linked to the basic problem?
* Do the treatment effects persist 6 months after the treatment has ended?

A prospective, non-inferiority randomised controlled study (RCT) with a number of (N=72) participants will be conducted to answer the study aims. A qualitative interview study will also be conducted to find out how the patients experience AA as an adjunctive therapy.

The participants will be randomised in two groups. The participants in group 1 will receive AA as an adjunctive therapy to TaU (i.e. individual counseling therapy, psycho therapy, pharmacological therapy) during 8 weeks. The add-on treatment will be administered at the treatment sessions with their caregiver (i.e. registered nurse, psychologist, curator), and at each session the participants receive 5 sterile stainless needles in each outer ear. The needling is standardised according to the NADA-protocol (10). The needles will remain in the outer ears for approximately 45 minutes, and will be removed by the care giver. Group 2, the control group, will receive TaU and will, just like group 1, have a follow-up after 8 weeks.

During the trial 12-15 participants from the AA group will be recruited to participate in an interview study. Semistructured interviews will be conducted after the 8 weeks intervention has finished. The questions are aimed to find out how the participants experienced the AA as an add-on treatment, and if AA was helpful to reduce symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria

* men and women aged 18 - 75
* diagnosis within the anxiety syndrome area (F. 41)
* post traumatic stress syndrome (PTSD) with mixed symptoms of anxiety and depression (F.309.28).

Exclusion Criteria

* psychotic symptoms
* increased risk for suicide
* intellectual impairment
* recent change- or start-up of pharmacological therapy
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory | Change from Baseline to end of treatment (8 weeks after baseline measurement) and change from baseline to 6 months after the end of treatment.
  A self-assessment scale to measure the prevalence of anxiety, worry and anxiety. Range of score is 20 to 80 in each subtest, the higher score indicate greater anxiety. The cutoff point is 39-40. STAI is the study's primary outcome measure.

SECONDARY OUTCOMES:
The Patient Health Questionnaire | Change from Baseline to end of treatment (8 weeks after baseline measurement) and change from baseline to 6 months after the end of treatment..
  A concise self-assessment scale for screening for actual depression and measuring the current symptom level of depression. Minimum score is 0 and maximum score is 27. The higher score indicate more severe depression. The cutoff points are 5, 10, 15 and 20 representing mild, moderate, moderately severe and severe levels of depressive symptoms.

OTHER OUTCOMES:
The Insomnia Severity Index | Change from Baseline to end of treatment (8 weeks after baseline measurement) and change from baseline to 6 months after the end of treatment.
  A self-assessment scale to measure the incidence of insomnia symptoms and the effect of initiated treatment. The total score ranges from 0 to 28, a higher score suggests more severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Lena U Bergdahl, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden